CLINICAL TRIAL: NCT07397520
Title: The Application of Intralesional 5-fluorouracil for the Management of Hypertrophic Facial Scars in the Periocular Region Resulting From Trauma and Surgical Procedures in Individuals Aged Over 18 Years
Acronym: AI5FMHFSPRFSOE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEI-2025/07/04
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Facial Scarring
Keywords: 5-FU; Fibrotic Scar; Facial Scarring

STUDY DESIGN:
Intervention Model Description: Intralesional administration of 5-fluorouracil will be conducted in the periocular scar. For the objective assessment of baseline status and subsequent facial skin changes, the validated Manchester Scar Scale will be used, which is a visual photonumeric scale for evaluating scar quality. This scale assesses six skin parameters, such as color, contour, distortion, texture, and brightness, assigning values from 1 to 4, with 1 indicating the best characteristic and 4 the least desirable.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intralesional administration of 5-fluorouracil will be conducted in the periocular scar group (Experimental): For the objective assessment of baseline status and subsequent facial skin changes, the validated Manchester Scar Scale will be used, which is a visual photonumeric scale for evaluating scar quality. This scale assesses six skin parameters, such as color, contour, distortion, texture, and brightness, assigning values from 1 to 4, with 1 indicating the best characteristic and 4 the least desirable.
  Interventions: Drug: Intralesional administration of 5-fluorouracil

INTERVENTIONS:
Drug: Intralesional administration of 5-fluorouracil — For the objective assessment of baseline status and subsequent facial skin changes, the validated Manchester Scar Scale will be used, which is a visual photonumeric scale for evaluating scar quality. This scale assesses six skin parameters, such as color, contour, distortion, texture, and brightness, assigning values from 1 to 4, with 1 indicating the best characteristic and 4 the least desirable

SUMMARY:
To determine the effectiveness of intralesional 5-fluorouracil in objectively reversing hypertrophic scars in the periocular region resulting from trauma or cosmetic surgery.

DETAILED DESCRIPTION:
During the initial visit, informed consent will be obtained and documented, alongside baseline photographs and measurements of the facial scar dimensions using a ruler. In the subsequent visits-second, third, fourth, and fifth-0.5 ml of intralesional 5-fluorouracil, diluted to 25 mg/ml, will be administered. Clinical photographs will be captured, and dimensions will be measured at each of these visits. A total of 0.5 ml of this solution will be injected weekly into the lesion to be treated, amounting to four doses over the course of one month.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants include male and female individuals over the age of 18 who possess a facial scar in the periocular region resulting from trauma or facial cosmetic surgery. Participants must voluntarily consent to partake in the study and have duly signed the requisite consent forms.

Exclusion Criteria:

* Exclusion criteria encompass the presence of local infections or inflammatory disorders, an allergy to 5-fluorouracil, pregnancy or breastfeeding, and any loss of control or follow-up during the study. Additionally, individuals experiencing local or systemic adverse reactions during the research are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in the size of facial hypertrophic scars | From enrollment to the end of treatment at 4 weeks
  To objectively assess baseline status and subsequent changes in facial skin, the validated photometric visual scale from Manchester, designed for evaluating scar quality, will be employed. This scale assesses six skin parameters, including coloration, contour, distortion, texture, and brightness, assigning values from 1 to 4, where 1 represents the most favorable characteristic and 4 the least desirable

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Oftalmologia F.A.P. Conde de Valenciana, I.A.P., Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From November to December 2026

REFERENCES:
- [Result] Browne RH. On the use of a pilot sample for sample size determination. Stat Med. 1995 Sep 15;14(17):1933-40. doi: 10.1002/sim.4780141709. PMID 8532986
- [Result] Leinonen M, Saikku P. Infections and atherosclerosis. Scand Cardiovasc J. 2000;34(1):12-20. doi: 10.1080/14017430050142341. PMID 10816055
- [Result] Tuan TL, Nichter LS. The molecular basis of keloid and hypertrophic scar formation. Mol Med Today. 1998 Jan;4(1):19-24. doi: 10.1016/S1357-4310(97)80541-2. PMID 9494966
- [Result] Slemp AE, Kirschner RE. Keloids and scars: a review of keloids and scars, their pathogenesis, risk factors, and management. Curr Opin Pediatr. 2006 Aug;18(4):396-402. doi: 10.1097/01.mop.0000236389.41462.ef. PMID 16914994
- [Result] Rabello FB, Souza CD, Farina Junior JA. Update on hypertrophic scar treatment. Clinics (Sao Paulo). 2014 Aug;69(8):565-73. doi: 10.6061/clinics/2014(08)11. PMID 25141117
- [Result] Pinedo HM, Peters GF. Fluorouracil: biochemistry and pharmacology. J Clin Oncol. 1988 Oct;6(10):1653-64. doi: 10.1200/JCO.1988.6.10.1653. PMID 3049954
- [Result] Ogawa R, Akaishi S, Kuribayashi S, Miyashita T. Keloids and Hypertrophic Scars Can Now Be Cured Completely: Recent Progress in Our Understanding of the Pathogenesis of Keloids and Hypertrophic Scars and the Most Promising Current Therapeutic Strategy. J Nippon Med Sch. 2016;83(2):46-53. doi: 10.1272/jnms.83.46. PMID 27180789
- [Result] Longley DB, Harkin DP, Johnston PG. 5-fluorouracil: mechanisms of action and clinical strategies. Nat Rev Cancer. 2003 May;3(5):330-8. doi: 10.1038/nrc1074. PMID 12724731
- [Result] Kim S, Woo YR, Cho SH, Lee JD, Kim HS. Clinical Efficacy of 5-Fluorouracil and Bleomycin in Dermatology. J Clin Med. 2024 Jan 6;13(2):335. doi: 10.3390/jcm13020335. PMID 38256469
- [Result] Lee HJ, Jang YJ. Recent Understandings of Biology, Prophylaxis and Treatment Strategies for Hypertrophic Scars and Keloids. Int J Mol Sci. 2018 Mar 2;19(3):711. doi: 10.3390/ijms19030711. PMID 29498630
- [Result] Ogawa R. Keloid and Hypertrophic Scars Are the Result of Chronic Inflammation in the Reticular Dermis. Int J Mol Sci. 2017 Mar 10;18(3):606. doi: 10.3390/ijms18030606. PMID 28287424
- [Result] Haurani MJ, Foreman K, Yang JJ, Siddiqui A. 5-Fluorouracil treatment of problematic scars. Plast Reconstr Surg. 2009 Jan;123(1):139-148. doi: 10.1097/PRS.0b013e3181904d1b. PMID 19116547
- [Result] Goldan O, Weissman O, Regev E, Haik J, Winkler E. Treatment of postdermabrasion facial hypertrophic and keloid scars with intralesional 5-Fluorouracil injections. Aesthetic Plast Surg. 2008 Mar;32(2):389-92. doi: 10.1007/s00266-007-9109-3. PMID 18185952
- [Result] Limandjaja GC, Niessen FB, Scheper RJ, Gibbs S. Hypertrophic scars and keloids: Overview of the evidence and practical guide for differentiating between these abnormal scars. Exp Dermatol. 2021 Jan;30(1):146-161. doi: 10.1111/exd.14121. Epub 2020 Jul 6. PMID 32479693
- [Result] Diasio RB, Harris BE. Clinical pharmacology of 5-fluorouracil. Clin Pharmacokinet. 1989 Apr;16(4):215-37. doi: 10.2165/00003088-198916040-00002. PMID 2656050
- [Result] Atiyeh BS. Nonsurgical management of hypertrophic scars: evidence-based therapies, standard practices, and emerging methods. Aesthetic Plast Surg. 2007 Sep-Oct;31(5):468-92; discussion 493-4. doi: 10.1007/s00266-006-0253-y. Epub 2007 Jun 18. PMID 17576505
- [Result] Ehrlich HP, Desmouliere A, Diegelmann RF, Cohen IK, Compton CC, Garner WL, Kapanci Y, Gabbiani G. Morphological and immunochemical differences between keloid and hypertrophic scar. Am J Pathol. 1994 Jul;145(1):105-13. PMID 8030742
- [Result] Jiang ZY, Liao XC, Liu MZ, Fu ZH, Min DH, Yu XT, Guo GH. Efficacy and Safety of Intralesional Triamcinolone Versus Combination of Triamcinolone with 5-Fluorouracil in the Treatment of Keloids and Hypertrophic Scars: A Systematic Review and Meta-analysis. Aesthetic Plast Surg. 2020 Oct;44(5):1859-1868. doi: 10.1007/s00266-020-01721-2. Epub 2020 Apr 27. PMID 32342167
- [Result] Shah VV, Aldahan AS, Mlacker S, Alsaidan M, Samarkandy S, Nouri K. 5-Fluorouracil in the Treatment of Keloids and Hypertrophic Scars: A Comprehensive Review of the Literature. Dermatol Ther (Heidelb). 2016 Jun;6(2):169-83. doi: 10.1007/s13555-016-0118-5. Epub 2016 Apr 22. PMID 27105629